CLINICAL TRIAL: NCT00651781
Title: A Phase I/II National, Open-label, Multicenter Study of Bortezomib (Velcade) in Combination With FLAG-IDA (VFLAG- IDA) in Patients With Relapsed or Refractory Acute Myeloid Leukemia (AML).
Brief Title: Velcaflagida in Relapsed or Refractary Acute Myeloid Leukemia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: PETHEMA Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Nº EudraCT: 2005-004370-24; IIS-VEL-EU-070/26866138CAN2015
Record Dates: First submitted 2008-03-31; First posted 2008-04-03 (Estimated); Last update posted 2013-02-28 (Estimated); Status verified 2013-02

CONDITIONS: Acute Myeloid Leukemia
Keywords: Acute Myeloid Leukemia; Relapsed; Refractory
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Recurrence | interventions — Bortezomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Phase I:3 dose levels Cytarabine (200 mg/m2- 500 mg/m2-1000 mg/m2) with scheme Flag-Ida in combination with Velcade until determinate the appropriate dose.
  Phase II:
  Fludarabine, Cytarabine and Idarubicin in combination with 2 times per week of Velcade administration. Each 28-day treatment, patients will be evaluated, and in absence of disease progression or unacceptable toxicity, patients will start second cycle with Bortezomib in monotherapy two times per week followed by a 10 days rest period. That is, patients who response with acceptable toxicity will receive the combined sequential scheme twice (as induction and consolidation).
  Interventions: Drug: Bortezomib

INTERVENTIONS:
Drug: Bortezomib — 2 times per week of Velcade administration.

SUMMARY:
The primary aim of this study is:

• To analyze the efficacy (in order to evaluate the response) of a sequential treatment scheme of Bortezomib in combination with Fludarabine,Cytarabine and Idarubicin continued with Bortezomib monotherapy for patients with relapsed or refractory AML ≥18 years old.

The safety aim of this study is:

• To evaluate the safety and tolerance of the sequential treatment scheme proposed with Bortezomib combined with Fludarabine, Cytarabine and Idarubicin and in monotherapy, measured on clinical toxicities and laboratory incidences.

The biological aim of this study is:

• To evaluate the Minimal Residual Disease (MRD)impact that will be monitored by multiparametric flow cytometry carried out at different moments during the treatment.

DETAILED DESCRIPTION:
Initially a phase I will be performed to determine the appropriate dose of Cytarabine to be used in Flag-Ida regimen in combination with Velcade; for that reason, first 9 patients will be distributed to 3 different cohorts with 3 patients in each cohort, which will be treated at each Cytarabine dose level (200 mg/m2-500 mg/m2-1000 mg/m2)in combination with the other drugs from Flag scheme and the fixed dose of Velcade at 1,3 mg/m2.

Once the appropriate Cytarabine dose is determined,the recruitment will be completed with 40 patients and evaluations and visits program will be realized in three periods: Pre-treatment, Treatment and Follow-up.

The Pre-treatment includes Screening and baseline visits. After providing informed consent, patients will be evaluated for study eligibility.

Eligible patients included in the study will receive the first cycle, which consist of Fludarabine, Cytarabine and Idarubicin in combination with 2 times per week of Velcade administration. Each 28-day treatment, patients will be evaluated, and in absence of disease progression or unacceptable toxicity, patients will start second cycle with Bortezomib in monotherapy two times per week followed by a 10 days rest period. That is, patients who response with acceptable toxicity will receive the combined sequential scheme twice (as induction and consolidation).

Patients will be evaluated the day 1 of each cycle,during the treatment period, in order to know the response before carrying on the treatment. Once the Treatment period is completed, patients will be evaluated during the Follow-up period, one monthly visit in year 1, and every 3 months for 3 next years. On each center criteria, autologous/allogeneic transplant can be planned depending on age and HLA identical sibling donor make it possible: it will be done following the sequential scheme (Velcade-Flag-Ida and Velcade in monotherapy); if the patient is not candidate for a transplant or has no donor, he/she will receive 2 sequential scheme.

Safety will be evaluated through all adverse events monitoring, physical exploration, vital signs, hematimetric and biochemical analysis. The treatment response will be evaluated using Cheson's standardized criteria, and MRD impact will be necessary evaluated the day 1 of each new cycle before to carry on the treatment.

ELIGIBILITY:
Inclusion Criteria:

* The patient must, according with investigator criteria,be able to comply with all the protocol requirements.
* The patient must sign voluntarily the informed consent before the performance of any study related procedure not part of usual medical care, with the knowledge that can leave the study the moment he/she wants, without prejudice to later medical care.
* Age ¡Ý 18 years old.
* Patient must be diagnosed with AML according World Health Organization (WHO)18 criteria (see Appendix 7).
* Patient with refractory AML after standard therapy, or relapsed AML after standard therapy or hematopoietic progenitors transplant (autologous or allogenic).
* Patient has a ECOG performance status <= 2 (see Appendix 5).
* Patient has the following laboratory values before Baseline visit:

  1. Platelet count ≥ 30000/mm3 (transfusion allowed), hemoglobin ≥ 8 g/dl (transfusion allowed) and absolute neutrophil count ≥ 0.750/mm3. Lower values are accepted if they are caused by bone marrow infiltration.
  2. Aspartate transaminase (AST): ≤ 2.5 x the upper limit of normal.
  3. Alanine transaminase (ALT): ≤ 2.5 x the upper limit of normal.
  4. Total bilirubin: ≤1.5 x the upper limit of normal.
  5. Serum creatinine value ≤ 2 mg/dl.
* Negative pregnant test for fertile females

Exclusion Criteria:

Prior Bortezomib therapy.

* Promyelocytic AML.
* Patient has > Grade 2 peripheral neuropathy within 14 days before enrollment.
* Fertile patient is not going to use a medical effective contraceptive method during the trial.
* Patient has received other investigational drugs within 30 days before enrollment.
* Patient is known to be seropositive for the human immunodeficiency virus (HIV), Hepatitis B surface antigen-positive or active hepatitis C infection.
* Patient had a myocardial infarction within 6 months of enrollment or has New York Heart Association (NYHA) Class III or IV, heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias,or electrocardiographic evidence of acute ischemia or active conduction system abnormalities.
* Patient is enrolled in another clinical research study and/or is receiving an investigational agent for any reason.
* Pregnant or breast-feeding women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2008-04; Primary Completion 2013-01 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Efficacy (in order to evaluate the response) of a sequential treatment scheme of Bortezomib in combination with Fludarabine,Cytarabine and Idarubicin continued with Bortezomib monotherapy for patients with relapsed or refractory AML ≥18 years old. | 1 year

SECONDARY OUTCOMES:
Evaluate the safety and tolerance of the sequential treatment scheme proposed with Bortezomib combined with Fludarabine, Cytarabine and Idarubicin and in monotherapy, measured on clinical toxicities and laboratory incidences | 1 year
Evaluate the Minimal Residual Disease (MRD)impact that will be monitored by multiparametric flow cytometry carried out at different moments during the treatment | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: San Miguel Jesús, Dr, Study Chair — PETHEMA Foundation
Locations (13):
- Spain (13):
  - Hospital Universitario de Salamanca, Salamanca, Salamanca
  - Hospital Juan Canalejo, A Coruña
  - Hospital Germans Trias I Pujol, Badalona
  - Hospital Clinic y Provincial de Barcelona, Barcelona
  - Hospital Santa Creu y Sant Pau.Barcelona, Barcelona
  - Hospital Vall d´hebron, Barcelona
  - Hospital 12 de Octubre, Madrid
  - Hospital Clínico San Carlos., Madrid
  - Hospital Ramón y Cajal. Madrid, Madrid
  - Hospital Morales Messeguer, Murcia
  - Hospital Central de Asturias, Oviedo
  - Hospital La Fe de Valencia, Valencia
  - Hospital Lozano Blesa, Zaragoza

REFERENCES:
- See also: Spanish association of Haematology — http://www.aehh.org